CLINICAL TRIAL: NCT01677754
Title: A Phase II, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Investigate the Efficacy and Safety of RO4602522 Added to Background Alzheimer's Disease Therapy in Patients With Moderate Severity Alzheimer's Disease
Brief Title: A Study of RO4602522 in Participants With Moderate Severity Alzheimer Disease on Background Alzheimer Disease Therapy
Acronym: MAyflOwer RoAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP28248; 2012-000943-29 (EudraCT Number)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — sembragiline; Donepezil; Memantine; Rivastigmine; Galantamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo as add-on to a background therapy of AChEI (donepezil, rivastigmine, or galantamine) alone or in combination with memantine.
  Interventions: Drug: Placebo; Drug: Donepezil; Drug: Memantine; Drug: Rivastigmine; Drug: Galantamine
- RO4602522 1 milligram (mg) (Experimental): Participants will receive RO4602522 1 mg as add-on to a background therapy of AChEI (donepezil, rivastigmine, or galantamine) alone or in combination with memantine.
  Interventions: Drug: RO4602522; Drug: Donepezil; Drug: Memantine; Drug: Rivastigmine; Drug: Galantamine
- RO4602522 5 mg (Experimental): Participants will receive RO4602522 5 mg as add-on to a background therapy of AChEI (donepezil, rivastigmine, or galantamine) alone or in combination with memantine.
  Interventions: Drug: RO4602522; Drug: Donepezil; Drug: Memantine; Drug: Rivastigmine; Drug: Galantamine

INTERVENTIONS:
Drug: RO4602522 — Participants will receive RO4602522 orally once daily for 12 months.
  Arms: RO4602522 1 milligram (mg); RO4602522 5 mg
Drug: Placebo — Participants will receive placebo for RO4602522 orally once daily for 12 months.
  Arms: Placebo
Drug: Donepezil — Stable dose as background medication
Drug: Memantine — Stable dose as background medication in combination with AChEIs
Drug: Rivastigmine — Stable dose as background medication
Drug: Galantamine — Stable dose as background medication

SUMMARY:
This Phase II, multicenter, randomized, double-blind, parallel-group, placebo-controlled study will evaluate the efficacy and safety of RO4602522 in participants with moderate severity Alzheimer's disease. Participants who are taking background therapy of acetylcholinesterase inhibitors (AChEI) alone or in combination with memantine for at least 4 months before screening will be randomized to receive either one of two doses of RO4602522 or placebo for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer disease, based on the National Institute of Neurological and Communicative Disorders and Stroke (NINCDS)/Alzheimer's Disease and Related Disorders Association (ADRDA) and Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV-TR) criteria
* Mini-Mental State Exam (MMSE) score at screening between 13 and 20, inclusive
* Body mass index (BMI) between 18 and 36 kilograms per square meter (kg/m^2) (inclusive) at screening
* Modified Hachinski Ischemia Score of less than or equal to (</=) 4
* Participants with Cornell Scale for Depression in Dementia (CSDD) scores </= 13 at screening
* Receiving treatment with donepezil, rivastigmine, galantamine or any AChEIs in combination with memantine for at least 4 months before screening, with their dose and formulation stabilized at least 3 months before screening. All formulation and dosages are allowed except donezepil 23 mg (alone or in combination)
* Females of childbearing potential must have a negative pregnancy test and must agree to use effective contraception
* Generally healthy and ambulatory or ambulatory-aided (i.e., walker or cane)
* Have a reliable caregiver or some other identified responsible person who has frequent contact with the participant

Exclusion Criteria:

* Any neurological or psychiatric condition that may occur currently or during the course of the study that can impair cognition or functioning that is not associated with Alzheimer's disease
* Background of mental retardation
* Uncontrolled behavioral symptoms incompatible with compliance or evaluability
* Alcohol and/or substance abuse or dependence (DSM-IV-TR) in the past 2 years, except nicotine use which is allowed. However, smokers treated with nicotine replacement therapy or bupropion are excluded
* Unstable or poorly controlled hypertension as assessed by the investigator regardless of whether or not the participant is taking antihypertensive medications
* Unstable or clinically significant cardiovascular disease that could be expected to progress, recur, or change during study period to such an extent that it could bias the assessment of the clinical or mental status of the participant
* Inadequate hepatic, renal or thyroid function
* Positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection
* Poorly controlled diabetes (glycosylated hemoglobin [HbA1c] greater than or equal to [>/=] 9 percent at screening)
* Requiring nursing home care. Participants living in assisted living facilities are allowed if a reliable caregiver is available (see inclusion criteria)
* Current treatment for Alzheimer's disease other than those listed in inclusion criteria
* Participation at any time in an active Alzheimer's disease vaccine study
* Participation in a passive Alzheimer's disease immunization study less than 1 year before screening except for a) participants where documented medical history indicate that they were randomized to the placebo group in these studies, b) participants treated with bapineuzumab where a 6-month exclusion period applies
* Recent (</= 12 weeks) or concomitant use of other Monoamine oxidase inhibitors (selective or not) including selegiline or rasagiline
* Antidepressant treatments are not allowed except for citalopram up to 20 mg daily, escitalopram up to 10 mg daily, paroxetine up to 30 mg daily, sertraline up to 100 mg daily and trazodone up to 100 mg daily. If treated with one of these antidepressants, the treatment should be present for at least 6 weeks at screening. All other antidepressants including other SSRIs, tricyclic antidepressants (TCAs), serotonin-norepinephrine reuptake inhibitors (SNRIs), St. John's wort and bupropion are excluded
* Anti-psychotic use within 4 weeks before screening is not permitted except risperidone up to 1.5 mg/day, quetiapine up to 100 milligrams per day (mg/day), olanzapine up to 5 mg/day, and aripiprazole up to 10 mg daily
* Anxiolytics/ hypnotics use is not permitted except for benzodiazepines of short or intermediate half-life for anxiety/sleeping disorders. Zolpidem (up to 5 mg/day), zopiclone (up to 7.5 mg/day), eszopiclone (up to 2 mg/day), trazodone (up to 50 mg/day, at bedtime) or zaleplon (up to 5 mg/day) is permitted for insomnia
* Anti-Parkinson's agents within 2 weeks before screening are not permitted
* Recent (less than 4 weeks prior to screening) or concomitant use of anticonvulsants
* Anticholinergics/ antihistaminics within 2 weeks before screening are not permitted, except i) if used episodically more than 3 days before the screening cognitive measurement, ii) non-sedating antihistaminic medications (without anticholinergic effects such as cetirizine) or peripheral anticholinergics without central anticholinergic effects (such as, trospium for the treatment of hyperactive bladder), which are permitted
* Recent (less than 1 week prior to screening) or concomitant use of opioid drugs (tramadol, methadone, propoxyphene, or meperidine), cyclobenzaprine and dextromethorphan
* Concomitant use of sympathomimetic drugs, including sympathomimetics in local anesthetics and ephedra supplements

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2012-10-24 (Actual); Primary Completion 2015-06-12 (Actual); Study Completion 2015-06-12 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Behavior Subscale (ADAS-Cog-11) Score at Month 12 | Baseline, Month 12

SECONDARY OUTCOMES:
Percentage of Participants Achieving Response, Defined as an Increase From Baseline of Less Than or Equal to (<=) 4 Points in ADAS-Cog-11 | Baseline, Month 12
Change From Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) Scale Score at Month 12 | Baseline, Month 12
Change From Baseline in Behavioral Pathology in Alzheimer's Disease Frequency-Weighted Severity Scale (BEHAVE-AD-FW) Score at Month 12 | Baseline, Month 12
Percentage of Participants With Worsening in BEHAVE-AD-FW Score | Baseline to Month 12
Change From Baseline in Apathy Evaluation Scale (AES) Score at 12 months | Baseline, Month 12
Change From Baseline in Alzheimer's Disease Cooperative Study Clinician Global Impression of Change (ADCS-CGIC) Scale Score at 12 months | Baseline, Month 12
Percentage of Participants With Worsening in ADCS-CGIC Score | Baseline to Month 12
Change From Baseline in Global Deterioration Scale (GDS) Score at 12 months | Baseline, Month 12
Change From Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) Score at 12 months | Baseline, Month 12
Percentage of Participants with Adverse Events | Baseline up to 13 months
Percentage of Participants with Change in Lens Opacity Grading | Baseline; Months 6, and 12
Percentage of Participants with Abnormal Visual Acuity Test Results | Baseline, Months 6, and 12
Change From Baseline in Michigan Neuropathy Screening Instrument Score | Baseline, Weeks 8, 18, 30, 44, 52, and at the last follow-up visit (12 weeks after last dose, up to 64 weeks)
Percentage of Participants Receiving Concomitant Medications | Baseline to 13 Months
Apparent Total Clearance of the Drug From Plasma After Administration of RO4602522 | Day -1, pre-dose (0 hour) on Days 14, 28, 84, 168, 252, and 364; 1 to 2 hour post dose on Days 14, 84, 252; 2-4 and 5-6 hours post dose on Days 28, 168, and 364
Apparent Volume of Distribution at Steady State after Administration of RO4602522 | Day -1, pre-dose (0 hour) on Days 14, 28, 84, 168, 252, and 364; 1 to 2 hour post dose on Days 14, 84, 252; 2-4 and 5-6 hours post dose on Days 28, 168, and 364
Area Under the Plasma Concentration-Time Curve of RO4602522 | Day -1, pre-dose (0 hour) on Days 14, 28, 84, 168, 252, and 364; 1 to 2 hour post dose on Days 14, 84, 252; 2-4 and 5-6 hours post dose on Days 28, 168, and 364
Maximum Plasma Concentration of RO4602522 | Day -1, pre-dose (0 hour) on Days 14, 28, 84, 168, 252, and 364; 1 to 2 hour post dose on Days 14, 84, 252; 2-4 and 5-6 hours post dose on Days 28, 168, and 364

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (142):
- United States (42):
  - Advanced Research Center, Inc.;In-Patient Unit, Anaheim, California
  - Neurology Center of North Orange County, Fullerton, California
  - Torrance Clinical Research, Lomita, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Neurological Research Inst, Santa Monica, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Meridien Research, Brooksville, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Neurologic Consultants, P.A., Fort Lauderdale, Florida
  - Galiz Research, LLC, Hialeah, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Compass Research East, LLC, Orlando, Florida
  - Comprehensive Clinical Development, Inc.- St. Petersburg, FL, St. Petersburg, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - iResearch Atlanta, Decatur, Georgia
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Alexian Brothers Neurosci Inst, Elk Grove Village, Illinois
  - Louisiana Research Associates, New Orleans, Louisiana
  - Booker, J. Gary, MD, APMC, Shreveport, Louisiana
  - Northern Michigan Neurology, Traverse City, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - New York University Medical Center;Child Study Center, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Radiant Research, Inc., Wyomissing, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Alzheimer's Research & Clinical Programs, Charleston, South Carolina
  - University of North Texas Health Science Center, Fort Worth, Texas
- Australia (9):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Central Coast Neurosciences Research, Erina, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Box Hill Hospital; Eastern Clinical Research Unit, Box Hill, Victoria
  - A.G.Mander Pty Ltd, Geelong, Victoria
  - Heidelberg Repatriation Hospital, Heidelberg, Victoria
  - Hollywood Specialist Centre, Nedlands, Western Australia
  - Neurodegenerative Disorders Research, Subiaco, Western Australia
- Canada (16):
  - The Medical Arts Health Research Group, Powell River, British Columbia
  - Vancouver Hospital - UBC Hospital Site, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - Capitol District Health Authority, Halilfax, Nova Scotia
  - True North Clinical Research Kentville, Kentville, Nova Scotia
  - Jbn Medical Diagnostic Services Inc., Burlington, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario
  - Ingram, Jennifer MD, Peterborough, Ontario
  - Toronto Memory Program (Neurology Research Inc.), Toronto, Ontario
  - The Centre for Memory and Aging, Toronto, Ontario
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - Recherches Neuro-Hippocame, Gatineau, Quebec
  - Clinique Neuro Rive-Sud, Greenfield Park, Quebec
  - Institut Universitaire de gériatrie de Sherbrooke; Service de gériatrie/pavillon Argyll, Sherbrooke, Quebec
  - McGill Univeristy; Douglas Mental Health University Institute; Neurological and Psychiatric, Verdun, Quebec
  - CHU de Quebec - Hôpital de l' Enfant Jésus, Québec
- Czechia (10):
  - NEUROHK s.r.o., Choceň
  - P-P Klinika, Kladno
  - Supervize s.r.o., Kutna Hora - Vnitrni Mesto
  - Clintrial,s.r.o., Prague
  - AD71 s.r.o., Prague
  - Psychiatry Trial s.r.o., Prague
  - Neurologicka ambulance, Prague
  - FORBELI s.r.o., Prague
  - Nemocnice Na Bulovce, Prague
  - Thomayerova nemocnice, Praha 4 - Krc
- France (12):
  - Centre Hospitalier de la côte Basque, Bayonne
  - Hopital Neurologique Pierre Wertheimer, Bron
  - Hopital Nord Laënnec - CHU Nantes, Nantes
  - Hopital Cimiez; CMRR, Nice
  - Hôpital Lariboisière, Paris
  - Groupe Hospitalier Sud - Hôpital Xavier Arnozan, Pessac
  - Hôpital Maison Blanche, Reims
  - CHU Rennes - Hopital Hôtel Dieu, Rennes
  - CHU Toulouse - La Grave, Toulouse
  - CHU Tours - Hôpital Bretonneau, Tours
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
  - Hopital des Charpennes, Villeurbanne
- Germany (5):
  - Gemeinschaftspraxis, Ellwangen
  - Henriettenstiftung Hannover, Hanover
  - ISPG - Institut fuer Studien zur Psychischen Gesundheit, Mannheim
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Zentrum f. Neurologisch- Psychiatrische Studien und Begutachtung, Siegen
- Italy (8):
  - Nuovo Ospedale Civile S.Agostino - Estense, Modena, Emilia-Romagna
  - Policlinico Universitario Agostino Gemelli; Farmacia, Rome, Lazio
  - Fondazione Santa Lucia IRCCS, Rome, Lazio
  - Umberto I Policlinico di Roma-Università di Roma La Sapienza, Rome, Lazio
  - Ente Ospedaliero Ospedali Galliera, Genoa, Liguria
  - Università degli Studi di Genova, Genoa, Liguria
  - Azienda Ospedaliero Universitaria Pisana; Uff. Sperim. Clin. U.O. Farmaceutica, Pisa, Tuscany
  - Università degli studi di Perugia, Perugia, Umbria
- Poland (9):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Specjal. Praktyka Lekarska; Prof. Grzegorz Opala, Katowice
  - Centrum Medyczne Dendryt, Katowice
  - NZOZ NEURO-KARD Ilkowski i Partnerzy Sp. Partn. Lek, Poznan
  - NZOZ Syntonia, Pruszcz Gdański
  - NZOZ Pro-Cordis Sopockie Centrum Bad. Kardiolog, Sopot
  - mMED Maciej Czarnecki, Warsaw
  - Instytut Psychiatrii i Neurologii, Warsaw
- South Korea (9):
  - Dong-A University Hospital, Busan
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Inha University Hospital; Pulmonary Medicine, Incheon
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (12):
  - Hospital General Universitario de Elche; Servicio de Farmacia, Elche, Alicante
  - Fundació ACE, BArcelon, Barcelona
  - Hospital General De Catalunya; Servicio de Neurologia, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Virgen del Puerto, Plasencia, Palencia
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - CAE Oroitu, Barakaldo, Vizcaya
  - Hospital Perpetuo Socorro, Servicio de Geriatria, Albacete
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Skanes Universitetssjukhus, Malmo Skanes Universitetssjukhus, Malmo, Malmo
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
- United Kingdom (8):
  - Cognitive Treatment & Research Unit, Crowborough
  - Ninewells Hospital, Dundee
  - Glasgow Memory Clinic, Glasgow
  - West London Cognitive Disorders Treatment and Research Unit; Lakeside Metal Health Unit, Isleworth
  - Institute of Psychiatry, London
  - Norwich Medical School, Norwich
  - Derriford Hospital, Plymouth
  - Memory Service North, Sheffield

REFERENCES:
- [Derived] Nave S, Doody RS, Boada M, Grimmer T, Savola JM, Delmar P, Pauly-Evers M, Nikolcheva T, Czech C, Borroni E, Ricci B, Dukart J, Mannino M, Carey T, Moran E, Gilaberte I, Muelhardt NM, Gerlach I, Santarelli L, Ostrowitzki S, Fontoura P. Sembragiline in Moderate Alzheimer's Disease: Results of a Randomized, Double-Blind, Placebo-Controlled Phase II Trial (MAyflOwer RoAD). J Alzheimers Dis. 2017;58(4):1217-1228. doi: 10.3233/JAD-161309. PMID 28550255